CLINICAL TRIAL: NCT05759663
Title: Randomized Controlled Trial of Minimal Incision Repair of Rectus Abdominis Diastasis Versus Repair of the Entire Diastasis
Brief Title: MIRRAD Versus Plication of Entire Diastasis Trial
Acronym: MIRRADRCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karlskoga Hospital (Unknown)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRRAD RCT
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Muscle Diastasis
Keywords: Postpartum; Diastasis of the Rectus Abdominis Muscles; Surgery
MeSH Terms: conditions — Diastasis, Muscle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIRRAD (Experimental): A 3 cm vertical incision is made above the umbilicus. The umbilicus is de-attached from the Linea alba so that Linea alba 5-7 cm above and 3-5cm below the umbilicus is exposed. The abdominal rectus muscle diastasis is then plicated with double layer barbed suture. The first suture line is over and over continuous suture and the second suture line continuous suture line. The umbilicus is then re-attached with a single stich .
  Interventions: Procedure: MIRRAD
- Plication of the entire diastasis arm (Active Comparator): A low transverse incision is made and the subcutaneous tissue along the Linea alba dissected. If there is any hernia present in the Linea alba, it is invaginated in a plicated suture line. The entire DRAM along the Linea alba is plicated with continuous sutures. Excessive skin and subcutaneous tissue along the incision is excised and the wound closed. The subcutaneous tissue is closed with interrupted 4-0 PDS stitches.
  Interventions: Procedure: Plication of the entire diastasis arm

INTERVENTIONS:
Procedure: MIRRAD — Repair of the diastasis with MIRRAD technique
  Arms: MIRRAD
Procedure: Plication of the entire diastasis arm — Plication of the entire diastasis
  Arms: Plication of the entire diastasis arm

SUMMARY:
Background Postpartum diastasis of the rectus abdominis muscles (DRAM) has gained increasing attention as a condition that may affect abdominal trunk function but that may be alleviated by surgery. Most techniques for surgical reconstruction of DRAM are, however, associated with high costs, postoperative pain and risk of surgical complications. The aim of the present study is to evaluate a Minimal Incision Repair of Rectus Abdominis Diastasis (MIRRAD) in a randomized controlled open label trial. Altogether 120 women will be included.

Population Postpartum women with DRAM of at least 2 cm.

Intervention Plication of Linea alba through a 3-5 centimeter long incision at the level of the umbilicus

Control Plication of the entire Linea alba through a low transverse incision.

Outcome Primary outcome: Abdominal function rated with the Disability Rating Index Secondary outcomes: Operative time, postoperative stay, surgical complications, sick leave, persisting pain orated with the Ventral Pain Hernia Questionnaire, cosmetic outcome rated with BODY-Q

Follow-up Follow-up one month and one year after surgery

Significance If the study shows that MIRRAD is equally effective as plication of the entire Linea alba one year after surgery, it may be introduced as a standard technique for DRAM. If it is not as effective, it may still be an alternative with advantages in terms of cost benefit and the possibility to perform it as a daycare procedure.

DETAILED DESCRIPTION:
Background

Diastasis of the rectus abdominis muscles (DRAM) is a well-known phenomenon that until recently has not attracted much attention. It may either develop in high age, often in combination with truncal obesity, or as the result of one or more pregnancies. Several studies, have, however, shown that post-partum DRAM may cause impaired abdominal trunk function, often combined with pelvic floor dysfunction and back pain. Studies have also shown that these problems can be reduced with surgery aimed at restoring the integrity of the Linea alba [1-3] The favorable outcomes in well-selected samples of post-partum women [4] have resulted in a widespread demand for broadened indications and that such surgery should be offered routinely to all post-partum women with abdominal trunk dysfunction. However, concerns have been raised regarding the costs and potential hazards from such a procedure for a condition that is associated with abdominal function impairment but no potential serious morbidity.

The surgical techniques for restoring abdominal wall function in women with postpartum DRAM are mainly based on experience from ventral hernia surgery. The aim of ventral hernia surgery is ultimately to reduce the hernia sac to the abdominal cavity and closing the hernia defect in a way that the risk of recurrences is minimized. This may either be carried with an open or endoscopic technique, and with or without mesh reinforcement. Most studies on DRAM surgery are thus focused on strengthening the entire Linea alba and minimizing the risk for recurrence. In case of restoring the abdominal trunk function in DRAM, however, the aim should rather be to prevent the rectus muscles from separating during tension and thereby leaving room for the midline bulge of the abdominal trunk and loss of tonus in the abdominal wall.

Surgery for DRAM should thus aimed at being cost-effective and atraumatic enough to be offered for a very large number of women in need of treatment for DRAM as well as to be safe enough to ensure that postoperative complications and early recurrences are not seen. For that purpose, we intend to evaluate a surgical technique that limits the surgical trauma and could be carried out in a large scale without need of great resources.

Study design

The study will be conducted as an open label randomized controlled trial where an established and evaluated technique, i.e., plication of the dilated part of Linea alba with open technique through a low transverse skin incision will be compared with MIRRAD. Before inclusion the woman should have undergone an organized training program without satisfying result. After consent has been given, the patient is randomized between MIRRAD or plication of the entire DRAM. Prior to surgery the patient undergoes examination by a physiotherapist and the Abdominal Trunk Function Protocol is completed. Regardless of allocation, the procedure is carried out under general anesthesia.

MIRRAD arm A 3 cm vertical incision is made above the umbilicus. The umbilicus is de-attached from the Linea alba so that Linea alba 5-7 cm above and 3-5cm below the umbilicus is exposed. The abdominal rectus muscle diastasis is then plicated with double layer barbed suture. The first suture line is over and over continuous suture and the second suture line continuous suture line. The umbilicus is then re-attached with a single stich . The skin is closed with continuous intradermal sutures.

Plication of the entire diastasis arm A low transverse incision is made and the subcutaneous tissue along the Linea alba dissected. If there is any hernia present in the Linea alba, it is invaginated in a plicated suture line. The entire DRAM along the Linea alba is plicated with continuous sutures. Excessive skin and subcutaneous tissue along the incision is excised and the wound closed. The subcutaneous tissue is closed with interrupted 4-0 PDS® stitches. The skin is closed with continuous intradermal sutures.

Follow-up Four hours after the procedure is completed the woman is requested to rate pain and nausea on VAS scales. All included women are invited to follow-up one month and one year after surgery. At the follow-up one month after surgery, postoperative complications, day of return to work are registered and the abdominal function is rated according to the Disability Rating Index of the Abdominal Trunk Function Protocol and persisting pain according to the Ventral Hernia Pain Questionnaire. At the one year postoperatively abdominal function is evaluated according to the Abdominal Trunk Function Protocol, persisting pain with Ventral Hernia Pain Questionnaire and cosmetic outcome with the belly contour items of the BODY-Q questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Women having undergone at least one pregnancy
* Age 20 - 50 years
* Minimum 2 cm diastasis of rectus abdominis muscle at the level of the umbilicus
* BMI < 30
* Treatment failure after six months of structured training

Exclusion Criteria:

* Nulliparous women
* Less than one year since last pregnancy
* Women who have not undergone structured training for at least six months
* Previous abdominal surgery through open midline incision
* Presence of excessive skin folds
* Future planned pregnancies

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Postpartum women
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal trunk function | One year
  Abdominal function assessed with Abdominal Trunk Function Protocol one year after surgery

SECONDARY OUTCOMES:
Operation time | Two hours
  Time required to complete the procedure
Postoperative pain 4 hours after surgery | Four hours
  Pain rated on a VAS scale
Postoperative nausea 4 hours after surgery | Four hours
  Nausea rated on a VAS scale
Time from surgery to discharge | Seven days
  Time from surgery to the moment when the patient is discharged
Surgical complications | Thirty days
  Complications related to the procedure rated according to Clavien-Dindo
Postoperative sick leave | Thirty days
  Time from surgery to full return to work
Postoperative seroma | Thirty days
  Subcutaneous confirmed at clinical examination 30 days postoperatively
Pain from abdominal wall | One year
  Pain from abdominal wall rated with VHPQ one month and one year after surgery
Abdominal Trunk function | One month
  Abdominal Trunk function assessed with Abdominal Trunk Function Protocol one month after surgery
Cosmetic satisfaction | One year
  Cosmetic outcome rated with BODY-Q one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sandblom, Ass prof, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Department of Surgery, Karloskoga Hospital, Karlskoga
  - Stockholm South General Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No